CLINICAL TRIAL: NCT03739216
Title: A Prospective, Multi-Center Registry of Subjects Treated With the ClariFix Cryotherapy Device
Brief Title: Registry of Subject Treated With ClariFix
Acronym: SNIF
Status: Completed | Type: Observational
Sponsor: Arrinex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-0004
Record Dates: First submitted 2018-10-03; First posted 2018-11-13 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Open label: Open label registry study of patients treated with the ClariFix device for chronic rhinitis.
  Interventions: Device: ClariFix

INTERVENTIONS:
Device: ClariFix — The ClariFix device is a handheld cryosurgical device which provides focal, controlled freezing to the target tissue.

SUMMARY:
A multi-center, prospective, non-randomized, observational registry to asses the results of the ClariFix(TM) device when used to ablate unwanted tissue in the nose of subjects with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to receive treatment with the ClariFix device in accordance with the ClariFix Instructions for Use.
* Participant is able to provide consent and willing to adhere to the study visit schedule.

Exclusion Criteria:

* Participant is scheduled to have additional treatment and/or procedures completed at the same time of treatment with the ClariFix device.
* Participant is scheduled to have additional nasal or sinus treatments and/or procedures completed within 3 months of treatment with the ClariFix device.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians and staff will invite patients receiving treatment with ClariFix device and who meet enrollment criteria to participate in the registry. Invited patients who provide informed consent will be enrolled into the registry. Baseline, treatment, and follow-up data will be collected at predetermined intervals.
Sampling Method: Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in nasal symptom severity | Follow-up visits at 6 weeks, 3, 6, 9, 12, 15, 18, 21, and 24 months post treatment
  Effectiveness will be assessed by the change from baseline in nasal symptoms using the TNSS (Total Nasal Symptom Score). The TNSS is a patient-reported assessment of 4 symptom scores for rhinorrhea (runny nose), nasal congestion, nasal itching, and sneezing. Each symptom is rated on a scale of 0 (none) to 3 (severe). The symptom scores are summed to give a total TNSS score that can range from 0 to 12.

SECONDARY OUTCOMES:
Patient-assessed improvement in nasal symptoms | Follow-up visits at 6 weeks, 3, 6, 9, 12, 15, 18, 21, and 24 months post treatment
  Percentage of participants reporting their change from baseline as minimally improved, much improved, or very much improved using the Patient Global Impression of Change (PGIC) assessment. The PGIC has patients evaluate their improvement over baseline on a scale from 1 (very much improved) to 7 (very much worse).
Clinician-assessed improvement in nasal symptoms | Follow-up visit at 3 months post treatment
  Percentage of clinicians reporting their participants change in nasal symptoms from baseline as minimally improved, much improved, or very much improved using the Clinical Global Impression - Improvement (CGI-I) assessment. The CGI-I has clinicians rate their patient's improvement over baseline on a scale from 1 (very much improved) to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Amber U Luong, MD, PhD, Principal Investigator — UT Health - The University of Texas
Locations (23):
- United States (23):
  - Del Rey Allergy & Sinus, Bakersfield, California
  - Del Rey Allergy & Sinus, Marina del Rey, California
  - Sacramento, Ear, Nose, and Throat, Roseville, California
  - UC Davis Dept of Otolaryngology, Sacramento, California
  - Breathe Clear Institutue, Torrance, California
  - Light ENT, Boynton Beach, Florida
  - Ear, Nose, and Throat Associates of South Florida, Plantation, Florida
  - North Georgia ENT, Cumming, Georgia
  - Chicago Nasal & Sinus, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Tandem Clinical Research, Marrero, Louisiana
  - Albany ENT & Allergy, Albany, New York
  - ENT & Allergy/Northwell Health, New York, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Piedmont ENT, Winston-Salem, North Carolina
  - Bethlehem ENT, Bethlehem, Pennsylvania
  - Texas Healthcare, Fort Worth, Texas
  - Collin County ENT, Frisco, Texas
  - UT Health, Houston, Texas
  - ENT Associates of Texas, McKinney, Texas
  - Ogden Clinic, Ogden, Utah
  - Metropolitan ENT, Alexandria, Virginia
  - Aurora Health System, Milwaukee, Wisconsin